CLINICAL TRIAL: NCT01864252
Title: The Effect of Remote Ischaemic Preconditioning and Glyceryl Trinitrate on Peri-operative Myocardial Injury in Cardiac Bypass Surgery Patients (ERIC-GTN Study)
Brief Title: Investigation Into the Role of GTN & RIPC in Cardiac Surgery
Acronym: ERIC-GTN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 120541
Record Dates: First submitted 2013-04-29; First posted 2013-05-29 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Myocardial Reperfusion Injury
MeSH Terms: conditions — Myocardial Reperfusion Injury | interventions — Saline Solution; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 Control (65 patients) (Sham Comparator): Sham Remote ischaemic preconditioning with IV normal saline 2-5ml/hour.
  Interventions: Drug: IV Normal saline
- Group 2 (65 patients) (Active Comparator): Patients administered a Remote Ischaemic preconditioning protocol (three-5 min cycles of simultaneous inflation to cuffs placed on upper arm and thigh) prior to surgery and IV normal saline 2-5 mL/h during surgery.
  Interventions: Other: Remote ischaemic preconditioning; Drug: IV Normal saline
- Group 3 GTN (65 patients): (Experimental): Patients administered sham simulated Remote Ischaemic Preconditioning protocol prior to surgery and IV Glyceryl Trinitrate 2-5ml/h during surgery.
  Interventions: Drug: IV Glyceryl trinitrate 2-5ml/h
- • Group 4 RIPC+GTN (65 patients): (Experimental): Patients administered Remote Ischaemic Preconditioning protocol and IV Glyceryl Trinitrate during surgery
  Interventions: Other: Remote ischaemic preconditioning; Drug: IV Glyceryl trinitrate 2-5ml/h

INTERVENTIONS:
Other: Remote ischaemic preconditioning — 3 cycles of 5 minutes to arm and legs
  Arms: Group 2 (65 patients); • Group 4 RIPC+GTN (65 patients):
Drug: IV Normal saline — Normal saline IV started prior to knife to skin at a rate of 2-5 mls/h and stopped just after weaning off bypass.
  Arms: Group 1 Control (65 patients); Group 2 (65 patients)
Drug: IV Glyceryl trinitrate 2-5ml/h — IV GTN given during surgery started prior to knife to skin and stopped after weaning off cardiopulmonary bypass.
  Arms: Group 3 GTN (65 patients):; • Group 4 RIPC+GTN (65 patients):

SUMMARY:
The purpose of this study is to determine whether Glyceryl Trinitrate (GTN) reduces injury to the heart during heart-lung bypass surgery in combination with the newer technique of remote ischaemic preconditioning (RIPC).

DETAILED DESCRIPTION:
Ischaemic heart disease is a leading cause of mortality in the western world. A number of patients undergo coronary artery bypass graft (CABG) surgery as treatment for ischaemic heart disease. With the rise of interventional procedures, patients who are coming to have CABG surgery are higher risk1. Remote ischaemic preconditioning (RIPC) has been shown to reduce perioperative myocardial injury (PMI) in patients having CABG even when cold blood cardioplegia or intermittent cross clamp fibrillation is used as cardioprotective measures. These patients have a general anaesthetic with multiple infusions including Glyceryl Trinitrate (GTN). The use of GTN in these patients is based on theoretical assumptions of coronary vasodilation pre operatively along with maintaining graft potency postoperatively. We intend to investigate the effect of GTN in patients undergoing cardiac surgery being subjected to RIPC in its role as a Nitric Oxide (NO) donor. Exogenous NO has been shown to be cardioprotective in animal models.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years all patients admitted for on- pump CABG and/or valve surgery
* Able to give consent

Exclusion Criteria:

* Allergies to excipients of IMP and placebo
* Chronic Renal failure (eGFR<30 ml/min/kg)
* Severe liver disease
* Peripheral arterial disease
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Troponin T area under the curve | 72 hours
  Troponin T area under the curve will be calculated using blood samples collected at 0,6,12,24,48 and 72 hours plotting it against time to calculated AUC.

SECONDARY OUTCOMES:
Inotrope/Vasopressor requirements peri-operatively | Post-operative day 1,2,3 and 4
  The inotrope score will be calculated as follows:
  Dosages (in μg/kg/min) of [Dopamine + Dobutamine] + [(Adrenaline + Noradrenaline + Isoproterenol + Isoproterenol) x 100] + [(Enoximone + Milrinone) x 15]
Ventilator dependence post operatively | Post-operative day 1,2,3 and 4
  The duration of endotracheal intubation will be noted in hours. Re-intubation rates will be calculated by noting down the number of patients requiring re-intubation and comparing this amongst the 4 groups.
Incidence of Acute Kidney Injury assessed using biomarkers | Post-operative day 1,2,3 and 4
  Serum creatinine levels will be noted in the first 3 days postoperatively. If a patient requires renal replacement therapy, this will be recorded and comparisons made amongst the groups. Hourly urine output and daily urine volumes for the duration of ITU stay will be recorded.
Length of ITU stay | Average 4 days
  A record of stay in days will be noted
Length of hospital stay | Average 14 days
  Duration of hospital stay will be recorded in days
Incidence of post-operative atrial fibrillation | Post-operative day 1,2,3 and 4
  Atrial fibrillation will be diagnosed using ECG. A record of the number of patients developing AF post operatively, the intervention used to treat it and whether or not the patient reverted to sinus rhythm prior to ITU discharge will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Derek Yellon, PhD DSc FRCP, Principal Investigator — The Hatter Cardiovascular Institute
Locations (1):
- The Heart Hospital, UCL Hospitals NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Hamarneh A, Sivaraman V, Bulluck H, Shanahan H, Kyle B, Ramlall M, Chung R, Jarvis C, Xenou M, Ariti C, Cordery R, Yellon DM, Hausenloy DJ. The Effect of Remote Ischemic Conditioning and Glyceryl Trinitrate on Perioperative Myocardial Injury in Cardiac Bypass Surgery Patients: Rationale and Design of the ERIC-GTN Study. Clin Cardiol. 2015 Nov;38(11):641-6. doi: 10.1002/clc.22445. Epub 2015 Sep 28. PMID 26412308